CLINICAL TRIAL: NCT02338687
Title: Low Dose Calcium Supplementation to Prevent Preeclampsia: a Cluster Randomized Study
Brief Title: Low Dose Calcium to Prevent Preeclampsia
Acronym: AMCAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: PPSUS (Programa Pesquisa para o SUS: gestão compartilhada em saúde) (Unknown); FAPEAM (Fundação de Amparo a Pesquisa do Estado do Amazonas) (Unknown); Universidade Federal do Amazonas (Other)
Responsible Party: Principal Investigator, Maria Regina Torloni, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 528759
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Pre-Eclampsia; Hypertension, Pregnancy-Induced; Dietary Calcium Deficiency
Keywords: Calcium; Dietary supplements; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Nutritional education; Diet therapy; Diet records; Hospitalization; Maternal mortality
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Maternal Death | interventions — Calcium; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: cluster randomized
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Active Comparator): Educational sessions
  Interventions: Behavioral: Educational sessions
- Education plus supplement (Experimental): Educational sessions and 500 mg calcium per day
  Interventions: Dietary Supplement: calcium; Behavioral: Educational sessions

INTERVENTIONS:
Dietary Supplement: calcium — one chewable tablet daily, at bedtime, containing 500 mg elemental calcium (1250 mg calcium carbonate)
  Arms: Education plus supplement
Behavioral: Educational sessions — Women will participate in at least 2 interactive group educational sessions lasting 30 minutes each. Session content: importance of calcium during pregnancy and how to modify their diets to include calcium-rich foods that are available locally
  Other Names: Dietary counseling

SUMMARY:
The purpose of this study is to assess, in pregnant women with calcium-poor diets, what is the effectiveness of low-dose (500 mg/day) calcium supplements associated with an educational intervention, compared to the educational intervention alone, in the prevention of preeclampsia and hypertensive disorders during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to understand verbal and visual instructions
* Gestational age 16 - 20 weeks
* Live fetus

Exclusion Criteria:

* Hyperparathyroidism or other contra-indication to calcium supplementation
* Gastrointestinal diseases or conditions that may interfere with calcium absorption (e.g. bariatric surgery, cancer, chronic colitis)
* Use of medications that may interfere with calcium absorption (e.g. corticosteroids, thiazides, thyroid hormones)
* Women already taking calcium supplements or daily antacids at recruitment

Ages: 10 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1040 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Preeclampsia | at 20-40 weeks of pregnancy
  New onset of hypertension plus proteinuria after 20 weeks of pregnancy
Hypertensive disorders of pregnancy | at 20-40 weeks of pregnancy
  New onset of hypertension, with or without proteinuria, after 20 weeks of pregnancy

SECONDARY OUTCOMES:
Mean change in dietary calcium intake | at 30-36 weeks of pregnancy
  At baseline, participants will provide a dietary record and again in the 3rd trimester. Changes in the mean dietary calcium intake will be calculated.
Hospital admission due to hypertension | at 20-40 weeks of pregnancy
  Admission (before labor) due to hypertension
Severe maternal morbidity | at 20-40 weeks of pregnancy
  Eclampsia or HELLP (Hemolysis, Elevated Liver Enzymes, Low Platelet) syndrome
Maternal mortality | starting at 20 weeks up to hospital discharge
  any cause maternal mortality
Gastrointestinal side effects of calcium | at 20-40 weeks of pregnancy
  incidence of flatulence, obstipation or other symptoms any time up to delivery
Maternal admission to Intensive Care Unit | at 20-40 weeks of pregnancy
  admission for any cause
Admission to Neonatal Intensive Care Unit | from delivery to infant discharge
  admission for any cause
Preterm birth | at 20-36 weeks
  Delivery before 37 weeks
Low birth weight | at 20-40 weeks
  Birth weight less than 2500 g
Small for gestational age infant | at 20-40 weeks
  Birth of an infant whose weight is below the 10th percentile for gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Maria Regina Torloni, MD, PhD, Study Chair — Sao Paulo Federal University
Locations (1):
- Universidade Federal do Amazonas, Manaus, Amazonas, Brazil